CLINICAL TRIAL: NCT02817256
Title: A Randomized Controlled Trial of Vitamin and Mineral Supplementation Post Bariatric Surgery: Sleeve Gastrectomy
Brief Title: Vitamin and Mineral Supplementation Post Bariatric Surgery
Acronym: RCTVMSSG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: United Arab Emirates University (Other)
Responsible Party: Principal Investigator, Juma Alkaabi, Professor, College of Medicine and Health Sciences, United Arab Emirates University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRD IRR 430#
Record Dates: First submitted 2016-06-19; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Complications of Other Bariatric Procedure
MeSH Terms: interventions — Vitamins; Minerals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A, 'vitamins and minerals' (Active Comparator): "Ergocalciferol , Vitamin B12, Calcium /D ", "Iron" or "Centrium".
  Ergocalciferol 300,000 IM - Every 3 months Oral Vitamin B12 tablets daily (500mcg) Calcium /D Tab 600-200mg Centrium -1 Tablet Daily
  Mineral:
  Iron preparation - Daily (47mg)
  Interventions: Dietary Supplement: Vitamins and Minerals
- Group B, 'vitamins and minerals' (Active Comparator): "Ergocalciferol , Vitamin B12, Calcium /D ", "Iron" or "Centrium".
  Centrium - 1 Tablet daily Ergocalciferol 50000 IU once every two weeks Vitamin B12 1000mcg IM every three months Calcium /D Tab 600-200mg
  Minerals:
  Iron preparation - Daily (47mg)
  Interventions: Dietary Supplement: Vitamins and Minerals

INTERVENTIONS:
Dietary Supplement: Vitamins and Minerals — Multivitamins and Minerals supplementation

SUMMARY:
Bariatric surgery is emerging as an essential treatment option for the management of obesity and its associated comorbidities. Many patients present for surgery have pre-existing low blood vitamin levels, thus all bariatric surgical procedures compromise nutrition to varying extents, and may present potential threat of micronutrient deficiencies. Therefore, long term nutritional monitoring and follow-ups are vital components of all bariatric surgical patients. However, there are no current standard practices in United Arab Emirates (UAE) for the biochemical monitoring and replacement of essential micronutrients in patients undergoing bariatric surgery particularly the most performed Sleeve Gastrectomy. Medical practice guidelines recommend nutritional care however, the dose and route of administration supplementation after surgery based on randomized controlled trials is not yet established. Till tow no scientific study has been performed on monitoring vitamins and minerals levels following bariatric surgery among UAE population. Therefore, present study is aimed to determine the dose and route of administration of vitamins and minerals in improving the micronutrient deficiencies post-operatively. Two standard different dosage forms (oral /parenteral) of vitamins and minerals will be given to the patients who had undergone sleeve gastrectomy at Tawam Hospital. The dosages of the supplementations are within the international recommendations and patients will be followed up closely for a period of one year. The effect of nutritional deficiencies on micronutrient level and quality of life (QOL) will be assessed. This will help the medical practitioners to prove the optimal possible nutrition for patients.

DETAILED DESCRIPTION:
The study will be conducted in Tawam Hospital where patients come for their routine bariatric surgery. A written informed consent will be taken from all the patients willing to participate in the study. Patients would be informed about the objectives / goals of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-60 years;
* No medical or psychiatric contraindications;
* BMI>35 kg/m2 with co-morbidities or BMI > 40 kg/m2 prior to the bariatric surgery.

Exclusion Criteria:

* • Documented severe micronutrient deficiency that require treatment

  * Documented poor compliance;
  * History of in concordance to medication;
  * Inflammatory bowel disease, malignant or debilitating medical conditions;
  * Known hemoglobinopathies or those diagnosed with pernicious anaemia;
  * Known history of kidney renal stones or history of hypercalcaemia;
  * Significant longstanding medical complications that affect micronutrient status;
  * Severe psychiatric illness;
  * Women who are lactating, pregnant or planning pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
monitor the levels of micronutrients of Iron | 1 year
  Change in micronutrients level of Iron

SECONDARY OUTCOMES:
monitor the levels of uric acid | 1year
  Change in level of uric acid
complications resulting from IM injections | 1 year
  Number of complications resulting from IM injections
monitor the levels of calcium | 1 year
  Change in level of calcium
monitor the levels of Vitamin A | 1 year
  Change in level of Vitamin A
monitor the levels of Vitamin D | 1 year
  Change in level of Vitamin D
monitor the levels of Serum folate | 1 year
  Change in level of Serum folate
monitor the levels of Vitamin B12 | 1 year
  Change in level of Vitamin B12
monitor the levels of Serum methyl malonate | 1 year
  Change in level of Serum methyl malonate

CONTACTS AND LOCATIONS:
Overall Officials: Salah Gariballa, MD, Study Chair — United Arab Emirates University
Locations (2):
- United Arab Emirates (2):
  - Faculty of Medicine and Health Sciences UAE University, Al Ain City, AB
  - Faculty of Medicine and Health Sciences, Al Ain City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gariballa S, Afandi B, Abuhaltem M, Yassin J, Habib H, Ibrahim W. Oxidative damage and inflammation in obese diabetic Emirati subjects supplemented with antioxidants and B-vitamins: a randomized placebo-controlled trail. Nutr Metab (Lond). 2013 Feb 4;10(1):21. doi: 10.1186/1743-7075-10-21. PMID 23379892
- [Result] Rhines SD, Heins JR. Pharmacotherapy for obesity and weight loss. S D Med. 2013 Nov;66(11):471, 473. No abstract available. PMID 24383264
- [Result] Bennett JM, Mehta S, Rhodes M. Surgery for morbid obesity. Postgrad Med J. 2007 Jan;83(975):8-15. doi: 10.1136/pgmj.2006.048868. PMID 17267672
- [Result] Coupaye M, Riviere P, Breuil MC, Castel B, Bogard C, Dupre T, Flamant M, Msika S, Ledoux S. Comparison of nutritional status during the first year after sleeve gastrectomy and Roux-en-Y gastric bypass. Obes Surg. 2014 Feb;24(2):276-83. doi: 10.1007/s11695-013-1089-6. PMID 24122661
- [Result] Batsis JA, Lopez-Jimenez F, Collazo-Clavell ML, Clark MM, Somers VK, Sarr MG. Quality of life after bariatric surgery: a population-based cohort study. Am J Med. 2009 Nov;122(11):1055.e1-1055.e10. doi: 10.1016/j.amjmed.2009.05.024. PMID 19854336
- [Result] Raoof M, Naslund I, Rask E, Karlsson J, Sundbom M, Edholm D, Karlsson FA, Svensson F, Szabo E. Health-Related Quality-of-Life (HRQoL) on an Average of 12 Years After Gastric Bypass Surgery. Obes Surg. 2015 Jul;25(7):1119-27. doi: 10.1007/s11695-014-1513-6. PMID 25566743
- [Result] Myers JA, Clifford JC, Sarker S, Primeau M, Doninger GL, Shayani V. Quality of life after laparoscopic adjustable gastric banding using the Baros and Moorehead-Ardelt Quality of Life Questionnaire II. JSLS. 2006 Oct-Dec;10(4):414-20. PMID 17575749
- [Result] Moize V, Andreu A, Flores L, Torres F, Ibarzabal A, Delgado S, Lacy A, Rodriguez L, Vidal J. Long-term dietary intake and nutritional deficiencies following sleeve gastrectomy or Roux-En-Y gastric bypass in a mediterranean population. J Acad Nutr Diet. 2013 Mar;113(3):400-410. doi: 10.1016/j.jand.2012.11.013. PMID 23438491
- [Result] Damms-Machado A, Friedrich A, Kramer KM, Stingel K, Meile T, Kuper MA, Konigsrainer A, Bischoff SC. Pre- and postoperative nutritional deficiencies in obese patients undergoing laparoscopic sleeve gastrectomy. Obes Surg. 2012 Jun;22(6):881-9. doi: 10.1007/s11695-012-0609-0. PMID 22403000
- [Result] Saif T, Strain GW, Dakin G, Gagner M, Costa R, Pomp A. Evaluation of nutrient status after laparoscopic sleeve gastrectomy 1, 3, and 5 years after surgery. Surg Obes Relat Dis. 2012 Sep-Oct;8(5):542-7. doi: 10.1016/j.soard.2012.01.013. Epub 2012 Feb 1. PMID 22398110
- [Result] Ruiz-Tovar J, Oller I, Tomas A, Llavero C, Arroyo A, Calero A, Martinez-Blasco A, Calpena R. Mid-term effects of sleeve gastrectomy on calcium metabolism parameters, vitamin D and parathormone (PTH) in morbid obese women. Obes Surg. 2012 May;22(5):797-801. doi: 10.1007/s11695-011-0582-z. PMID 22179702
- [Result] Gehrer S, Kern B, Peters T, Christoffel-Courtin C, Peterli R. Fewer nutrient deficiencies after laparoscopic sleeve gastrectomy (LSG) than after laparoscopic Roux-Y-gastric bypass (LRYGB)-a prospective study. Obes Surg. 2010 Apr;20(4):447-53. doi: 10.1007/s11695-009-0068-4. Epub 2010 Jan 26. PMID 20101473
- [Result] Majumder S, Soriano J, Louie Cruz A, Dasanu CA. Vitamin B12 deficiency in patients undergoing bariatric surgery: preventive strategies and key recommendations. Surg Obes Relat Dis. 2013 Nov-Dec;9(6):1013-9. doi: 10.1016/j.soard.2013.04.017. Epub 2013 May 24. PMID 24091055
- [Result] Pech N, Meyer F, Lippert H, Manger T, Stroh C. Complications and nutrient deficiencies two years after sleeve gastrectomy. BMC Surg. 2012 Jul 5;12:13. doi: 10.1186/1471-2482-12-13. PMID 22765843
- [Result] Eltweri AM, Bowrey DJ, Sutton CD, Graham L, Williams RN. An audit to determine if vitamin b12 supplementation is necessary after sleeve gastrectomy. Springerplus. 2013 May 10;2(1):218. doi: 10.1186/2193-1801-2-218. Print 2013 Dec. PMID 23741650
- [Result] Ruz M, Carrasco F, Rojas P, Codoceo J, Inostroza J, Basfi-Fer K, Valencia A, Csendes A, Papapietro K, Pizarro F, Olivares M, Westcott JL, Hambidge KM, Krebs NF. Heme- and nonheme-iron absorption and iron status 12 mo after sleeve gastrectomy and Roux-en-Y gastric bypass in morbidly obese women. Am J Clin Nutr. 2012 Oct;96(4):810-7. doi: 10.3945/ajcn.112.039255. Epub 2012 Sep 5. PMID 22952172
- [Result] Snyder-Marlow G, Taylor D, Lenhard MJ. Nutrition care for patients undergoing laparoscopic sleeve gastrectomy for weight loss. J Am Diet Assoc. 2010 Apr;110(4):600-7. doi: 10.1016/j.jada.2009.12.022. PMID 20338286
- [Result] Coupaye M, Breuil MC, Riviere P, Castel B, Bogard C, Dupre T, Msika S, Ledoux S. Serum vitamin D increases with weight loss in obese subjects 6 months after Roux-en-Y gastric bypass. Obes Surg. 2013 Apr;23(4):486-93. doi: 10.1007/s11695-012-0813-y. PMID 23150206
- [Result] Buchwald H, Oien DM. Metabolic/bariatric surgery worldwide 2011. Obes Surg. 2013 Apr;23(4):427-36. doi: 10.1007/s11695-012-0864-0. PMID 23338049
- [Result] Davies DJ, Baxter JM, Baxter JN. Nutritional deficiencies after bariatric surgery. Obes Surg. 2007 Sep;17(9):1150-8. doi: 10.1007/s11695-007-9208-x. PMID 18074487
- [Result] Rhode BM, Arseneau P, Cooper BA, Katz M, Gilfix BM, MacLean LD. Vitamin B-12 deficiency after gastric surgery for obesity. Am J Clin Nutr. 1996 Jan;63(1):103-9. doi: 10.1093/ajcn/63.1.103. PMID 8604656
- [Result] Sanchez-Hernandez J, Ybarra J, Gich I, De Leiva A, Rius X, Rodriguez-Espinosa J, Perez A. Effects of bariatric surgery on vitamin D status and secondary hyperparathyroidism: a prospective study. Obes Surg. 2005 Nov-Dec;15(10):1389-95. doi: 10.1381/096089205774859182. PMID 16354517
- [Result] Nimeri A, Mohamed A, El Hassan E, McKenna K, Turrin NP, Al Hadad M, Dehni N. Are results of bariatric surgery different in the Middle East? Early experience of an international bariatric surgery program and an ACS NSQIP outcomes comparison. J Am Coll Surg. 2013 Jun;216(6):1082-8. doi: 10.1016/j.jamcollsurg.2013.01.063. Epub 2013 Apr 23. PMID 23619317
- [Result] Heber D, Greenway FL, Kaplan LM, Livingston E, Salvador J, Still C; Endocrine Society. Endocrine and nutritional management of the post-bariatric surgery patient: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2010 Nov;95(11):4823-43. doi: 10.1210/jc.2009-2128. PMID 21051578
- [Result] Isom KA, Andromalos L, Ariagno M, Hartman K, Mogensen KM, Stephanides K, Shikora S. Nutrition and metabolic support recommendations for the bariatric patient. Nutr Clin Pract. 2014 Dec;29(6):718-39. doi: 10.1177/0884533614552850. Epub 2014 Oct 6. PMID 25288251
- [Result] Gudzune KA, Huizinga MM, Chang HY, Asamoah V, Gadgil M, Clark JM. Screening and diagnosis of micronutrient deficiencies before and after bariatric surgery. Obes Surg. 2013 Oct;23(10):1581-9. doi: 10.1007/s11695-013-0919-x. PMID 23515975